CLINICAL TRIAL: NCT03829878
Title: A Randomized Double-Blind Placebo Controlled Cross-Over Study of CP101 (Full-Spectrum Microbiota®) in Children With Autism Spectrum Disorder and Associated Gastrointestinal Symptoms
Brief Title: Efficacy, Safety, and Tolerability Study of Oral Full-Spectrum MicrobiotaTM (CP101) in Subjects With Autism Spectrum Disorder and Associated GI Symptoms (SPROUT)
Acronym: SPROUT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study not started
Sponsor: Finch Research and Development LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP101-ASD-203
Record Dates: First submitted 2019-01-28; First posted 2019-02-04 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Autism Spectrum Disorder; Autism; ASD; Autistic Thinking; Autistic Behavior; Finch; FMT; Fecal Microbiota Transplant; CP101; SPROUT; Fecal Transplant
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Child Development Disorders, Pervasive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CP101 (Experimental): CP101 (Full Spectrum Microbiota) Capsule
  Interventions: Drug: CP101
- Placebo (Placebo Comparator): Placebo for CP101
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CP101 — Orally administered donor derived full spectrum microbiota
  Other Names: FSM
  Arms: CP101
Drug: Placebo — Placebo for CP101
  Arms: Placebo

SUMMARY:
Adolescent autism spectrum disorder subjects with associated GI symptoms will be randomized to receive oral dosing of CP101 capsules in Treatment Group I or matching placebo capsules in Treatment Group II. The purpose of this study is to demonstrate the safety and effectiveness of CP101 in subjects with ASD and associated GI symptoms.

DETAILED DESCRIPTION:
This is a Randomized Double-Blind Placebo Controlled Study of CP101 (Full-Spectrum Microbiota®) in Children with Autism Spectrum Disorder and Associated Gastrointestinal Symptoms

ELIGIBILITY:
Inclusion Criteria:

* Male or Female ages 5 to 17
* Diagnosis of ASD by health care provider
* CARS-2 score ≥35 by the study evaluator
* 1 year history of chronic abnormal bowel function with/without GI symptoms
* GSRS/Constipation sub-score ≥3.0, or/and GSRS/diarrhea sub-score ≥3.0, during Screening

Exclusion Criteria:

* Inability to ingest intact capsules.
* Change or anticipated change of prescription medications and/or nutrition supplement and/or therapy to treat ASD symptoms
* Prior history, evidence, or diagnosis of inflammatory bowel disease or chronic autoimmune GI disease
* Below 5th percentile for weight on Centers for Disease Control and Prevention (CDC) growth chart based on age
* History of fecal microbiota transplantation (FMT) for any condition, regardless of route of administration within 12 months of Screening, or plan to undergo during the study
* History of epilepsy or any other seizure (except febrile seizure) disorder.
* Enrollment in any other investigational drug or device study within 8 weeks prior to investigational study medication (CP101/placebo) administration or within 5 half-lives of the last dose of the previous investigational compound, whichever is longer.
* Major intra-abdominal surgery within the past 60 days prior to Screening (excluding appendectomy or cholecystectomy) and/or planned invasive surgery/hospitalization during the study.
* Use of systemic antibiotics, systemic antiviral, or systemic antifungal (non-topical) for any condition during 8 weeks prior to Screening, or any anticipated use of above for any condition (e.g., frequent otitis media requiring antibiotics) before EOT (Week 24).
* Recent change or anticipated change of non-dietary probiotics.
* Any clinically significant condition that would jeopardize the safety or rights of the subject, or would confound the results of the study, in the opinion of the Principal Investigator.
* Clinically significant laboratory abnormalities at Screening at the discretion of the Principal Investigator.
* Pregnant, breast-feeding, or positive pregnancy test at Screening (for females of child-bearing potential) or for sexually active subjects (as determined by the Principal Investigator), who refuses to practice an acceptable form of birth control for the duration of the study.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Childhoood Autism Rating Scales-2 (CARS-2) | 24 weeks
  Two 15-item rating scales completed by the clinician (each designed for a different population); and an unscored Parent/Caregiver Questionnaire

SECONDARY OUTCOMES:
Aberrant Behavior Checklist-2 (ABC-2) | 55 weeks
  Scoring scale range from 1-3 for a 58 question, 5 behavior category assessments. All categories summed for individual total scores (7-48). Individual total scores determine severity (the higher, the more severe).
Social Responsiveness Scale-2 (SRS-2) | 55 weeks
  Total Score; Scores for 5 Treatment Subscales; Scores for 2 DSM-5 Compatible Subscales
Parent Global Impressions-III (PGI-III) | 55 weeks
  19 question assessment evaluating parent observations from "much worse" to "much better".
Gastrointestinal Symptom Rating Scale (GSRS) | 55 weeks
  Contains 15 items, uses a seven-graded Likert scale, where 1 represents the most positive option and 7 the most negative one.
Gastrointestinal Stool & Symptom Questionnaire for Autism (GSSQA) | 55 weeks
  17 item assessment evaluating GI symptoms on a scale from "Not at all" to "Almost always".
Reynolds Intellectual Assessment Scales-2-Nonverbal (RIAS-2-NV) | 55 weeks
  IQ test with 8 sub-categories. Scores from each category summed, then indexed
Autism Diagnostic Interview-Revised (ADI-R) | 55 weeks
  The ADI-R provides a diagnostic algorithm for autism as described in both the ICD-10 and DSM-IV. The instrument focuses on behavior in three main areas: qualities of reciprocal social interaction; communication and language; and restricted and repetitive, stereotyped interests and behaviors.

IPD SHARING:
Plan to Share IPD: No